CLINICAL TRIAL: NCT05071157
Title: Study of the Effects of Adolescent Weight Disorders (Obesity, Anorexia Nervosa) on Heart Function
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RBHP 2018 PAYSAL; 2018-A01907-48 (Other: 2018-A01907-48)
Record Dates: First submitted 2021-09-14; First posted 2021-10-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Anorexia Nervosa; Obesity
Keywords: cardiac function; adolescent; obesity; speckle tracking echocardiography; anorexia nervosa; metabolomic
MeSH Terms: conditions — Anorexia Nervosa; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for inflammatory factors (CRP, sedimentary rate, metabolomic)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- anorexia nervosa: girls between 12 and 18 years old with behavioral eating disorder characterized by a drastic reduction in intakes resulting in weight loss and a BMI ≤ 17.5 kg / m2. Anorexia can be restrictive pure or associated with bulimia
  Interventions: Behavioral: echocardiography
- obesity: girls between 12 and 18 years old with a BMI projecting ≥ 30 kg / m2 at the age of 18 (IOTF C30).
  Interventions: Behavioral: echocardiography
- normal weight: girls between 12 and 18 years old without BMI abnormality, without eating disorders, without serious medical pathology
  Interventions: Behavioral: echocardiography

INTERVENTIONS:
Behavioral: echocardiography — * speckle tracking echocardiography
  * evaluation of cardiac variability by recording heart rate as several hours (POLAR watch)
  * bioimpedance
  * blood test for biological assays (metabolomic analysis)

SUMMARY:
The study aims to better understand the functioning of the heart of children and adolescents with anorexia nervosa or obesity, compared to the heart function of control subject. This project seeks to find out if a weight disorder affects the heart and whether a systematic cardiac assessment with appropriate management is then to be considered.

To meet this objective, several analyzes are planned including a speckle tracking echocardiography, allowing a non-invasive study of myocardial deformations.

The hypothesis is that two opposite weight disorders (anorexia nervosa and obesity) lead to similar complications: inflammation, fibrosis altering the myocardial structure and therefore its contractility. Both systolic and diastolic dysfunction appear. Investigator hypothesize that the determinants of this dysfunction involve part of the alteration of body mass, and partly qualitative alterations specific to each pathology.

DETAILED DESCRIPTION:
The main objective is to evaluate the cardiac dysfunctions through the study of myocardial deformities in anorexic and obese adolescents, in comparison with controls. The choice of a pediatric population is explained by the probable precocity of the cardiac repercussions of these weight disorders. The desire to bring together in the same study two opposite weight disorders is because a certain number of complications are common to both: repercussions on the cardiac mass, presence of chronic systemic inflammation, and fibrosis. Comparison to normo-weighted healthy subjects will make it possible to determine whether certain alterations are directly attributable to body composition (in the case of a continuum of a parameter between the three groups) or, on the contrary, independent of body composition.

The search for the mechanisms at the origin of these alterations represents our secondary objective. For this, a correlation of the cardiac parameters with several factors such as: duration and severity of disorders, body composition, heart mass, presence of myocardial fibrosis, epicardial fat level, sympatho-vagal balance (by the cardiac variability), systemic inflammatory profile and potential pathways signaling involved (metabolomic analysis) will be carried out. All these parameters may impact cardiac function.

Adolescent girls participating in the study will benefit from a clinical examination with fat / lean body mass measurement by impedance, assessment of heart rate variability, blood test (inflammation marker, metabolomic analysis) and ultrasound heart. Thus, screening for heart disease, and more generally complications of their pathology, will be performed.

This project is important to answer the question of the necessity or not of a systematic cardiac assessment in these adolescents and the setting up of an adapted care

ELIGIBILITY:
Inclusion Criteria:

* girls between 12 and 18, affiliated to a social security
* with behavioral eating disorder characterized by a drastic reduction in intakes resulting in weight loss and a BMI ≤ 17.5 kg / m2. Anorexia can be restrictive pure or associated with bulimia
* or, with a BMI projecting ≥ 30 kg / m2 at the age of 18 (IOTF C30)
* or, without BMI abnormality, without eating disorders, without serious medical pathology

Exclusion Criteria:

* for anorexics, uncorrected nutritional deficiency
* for the obese, secondary obesity
* for all, inability to provide informed consent, pregnancy or breastfeeding, heart disease, high blood pressure, sleep apnea syndrome, dyslipidemia, diabetes, chronic pathology including inflammatory.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: girls between 12 and 18 with or without weight disorders
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
systolic global longitudinal strain | at inclusion
  echocardiographic parameter of myocardial deformation: index of myocardial systolic function in percent

SECONDARY OUTCOMES:
heart rate variability | at inclusion during first night
  holter measurement of standard deviation of all intervals between heart beat(SDNN) in ms
body composition | at inclusion
  fat mass and lean mass in percent
cardiac blood markers | at inclusion
  blood sampling: N-Terminal-proBNP in ng/L
inflammation blood markers | at inclusion
  blood sampling: CRP in mg/L
hormonal blood markers | at inclusion
  blood sampling: oestradiol in pg/ml
blood hemoglobin | at inclusion
  blood sampling: in g/L
ionogram blood markers | at inclusion
  blood sampling: blood potassium in mmol/l
heart rhythm and conduction | at inclusion
  electrocardiogram to determine ECG QT Interval

CONTACTS AND LOCATIONS:
Overall Officials: Justine Paysal, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France